CLINICAL TRIAL: NCT04852042
Title: Digital Health Supported Weight Management Intervention Delivered by Community Health Workers Among Public Housing Residents
Brief Title: Digital Health Weight Management Among Public Housing Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-41590; 1R01CA238335-01A1 (NIH)
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Weight Change, Body; Obesity
Keywords: Community health workers; Public housing residents; Behavioral interventions; Healthy eating; Physical activity
MeSH Terms: conditions — Body Weight Changes; Obesity; Motor Activity | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- mHealth Group (Experimental): 12 month text messaging program about diet and physical activity behavioral goals
  Interventions: Behavioral: mHealth
- mHealth+Community Health Worker (CHW) support (Experimental): same as mHealth group + monthly behavioral phone counseling by a CHW
  Interventions: Behavioral: mHealth; Behavioral: CHW support
- Control group (No Intervention): Assessments only

INTERVENTIONS:
Behavioral: mHealth — Participants will receive 2-3 text messages daily. The messages will include information to promote healthy eating and physical activity.
  Arms: mHealth Group; mHealth+Community Health Worker (CHW) support
Behavioral: CHW support — The CHW will provide behavioral counseling to participants guided by a study website related to their healthy eating and physical activity goals.
  Arms: mHealth+Community Health Worker (CHW) support

SUMMARY:
This research will test the efficacy of a weight management intervention through a three-group randomized trial: mHealth only, mHealth+Community Health Worker (CHW) support, versus control group, among residents of Boston's public housing developments. The mHealth group consists of a 1-year text messaging program to promote diet and physical activity behavior changes and the CHW support consists of monthly phone counseling delivered by a CHW to support the text messaging program. Our hypothesis is that the mHealth+CHW group will be more effective in bringing about weight loss compared to mHealth alone or the assessment only control group. The findings are expected to inform future health promotion efforts among residents in public housing developments.

ELIGIBILITY:
Inclusion Criteria:

* Current resident of Boston public housing development
* No plans to move within the next 6 months and no plan on leaving the country for more than 2 months over the next year
* Able to read and speak in English or Spanish
* Has cell phone with a plan that allows for unlimited text messages
* Willing to wear a device to track physical activity during assessment periods

Exclusion Criteria:

* Currently enrolled in a comprehensive weight loss program or a research study about weight that is incompatible with study participation
* Currently on a medically prescribed diet or fast that is incompatible with study participation
* Currently has a diagnosis of bipolar disorder, mania, manic-depressive disorder, schizophrenia, or psychosis and is not on any medications to treat the condition
* Precontemplation stage of change for making healthy eating or physical activity changes
* Pregnancy
* Medical contraindications to physical activity. Self-reported presence of any of the following:

  * Can not walk without help from someone else
  * Regularly needs to use the following special equipment to walk or get around: wheelchair, scooter, walker, or extra oxygen
  * Gets short of breath even when using special equipment at a very low level of physical activity such as walking around the home, making a bed, or taking a bath
  * Advised by a healthcare professional not to exercise and or if diagnosed with a bone or joint problem, it could get worse.
  * Frequently gets pains in the heart or chest
  * Had a heart attack in the past 6 months
  * Often feels faint or has spells of severe dizziness
  * Has very high blood pressure that is often over 175 or the bottom blood pressure number is often over 110
  * Has a good physical reason not to follow an activity program even if they wanted to

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2025-08-07 (Actual); Study Completion 2025-08-11 (Actual)

PRIMARY OUTCOMES:
Change in Weight at 12-month follow up | Baseline, 12-month follow up
  Weight will be objectively measured by study staff using standard procedures using an accurate electronic scale designed for portable use measured to the nearest 1/10th reading.

SECONDARY OUTCOMES:
Change in Weight at 6-month follow up | Baseline, 6-month follow up
  Weight will be objectively measured by study staff using standard procedures using an accurate electronic scale designed for portable use measured to the nearest 1/10th reading.
Diet behavior | Baseline, 6-month follow up, 12-month follow up
  Diet (for example: fruits & vegetables, whole grains, lean meats, and sugary beverages) will be measured via unannounced 24-hour recalls, one per person per assessment period. Other diet behaviors (for example: breakfast consumption) will be measured via questions on standardized surveys.
Physical activity behavior | Baseline, 6-month follow up, 12-month follow up
  Physical activity will be objectively measured via Actigraph 3tx accelerometers worn by participants for 7 days (minimum of 4 days) to assess time spent in light-to-moderate-to-vigorous physical activity.
Psycho-social variables | Baseline, 6-month follow up, 12-month follow up
  Psycho-social variables (for example: Self-efficacy, motivation, outcome expectations, depressive symptoms, sleep, social support) will be evaluated for change over the intervention period and whether they moderate the intervention effect on weight.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Quintiliani, PhD, Principal Investigator — Tufts Medical Center; Ziming Xuan, ScD, Principal Investigator — BU School of Public Health, Community Health Services
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Solar C, Nansubuga A, Murillo J, Ranker L, Borrelli B, Bowen DJ, Xuan Z, Kane J, Werntz S, Crouter SE, Quintiliani LM. Mobile health plus community health worker support for weight management among public housing residents (Path to Health): A randomized controlled trial protocol. Contemp Clin Trials. 2022 Aug;119:106836. doi: 10.1016/j.cct.2022.106836. Epub 2022 Jun 18. PMID 35724842